CLINICAL TRIAL: NCT05155137
Title: Polypill and RiscOMeter to Prevent StrOke and CogniTive ImpairmEnt in Primary Health Care
Brief Title: Polypill and RiscOMeter to Prevent StrOke and CogniTive ImpairmEnt (PROMOTE)
Acronym: PROMOTE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Moinhos de Vento (Other)
Collaborators: Ministry of Health, Brazil (Other Government); World Stroke Organization (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 41456820.6.1001.5330
Record Dates: First submitted 2021-11-30; First posted 2021-12-13 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Stroke; Cognitive Decline
Keywords: stroke; cognitive decline; prevention; polypill; stroke riskometer; primary care
MeSH Terms: conditions — Stroke; Cognitive Dysfunction | interventions — Pharmaceutical Preparations; Valsartan; Amlodipine; Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: Phase III, prospective, placebo-controlled randomized clinical trial involving 8,518 individuals in 80 Primary Care Health Units. Participants will be randomized into four groups: 1) Polypill (valsartan 80 mg, amlodipine 5 mg, and rosuvastatin 10 mg) + Stroke Riskometer, 2) Placebo + Stroke Riskometer, 3) Polypill + Usual care, and 4) Placebo + Usual care.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigator and patient will be blinded for polypill or placebo and the outcomes evaluator will be blinded for the treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Polypill + Stroke Riskometer (Experimental): Participants will be randomized to use the active polypill (valsartan 80 mg, amlodipine 5 mg, and rosuvastatin 10 mg) and to use the Stroke Riskometer for lifestyle modification
  Interventions: Drug: Drug Capsule (Valsartan + Amlodipine + Rosuvastatin); Behavioral: Stroke Riskometer
- Placebo + Stroke Riskometer (Placebo Comparator): Participants will be randomized to use placebo polypill and to use the Stroke Riskometer for lifestyle modification
  Interventions: Behavioral: Stroke Riskometer
- Polypill + No Stroke Riskometer (Usual care) (Experimental): Participants will be randomized to use the active polypill (valsartan 80 mg, amlodipine 5 mg, and rosuvastatin 10 mg) and will not use the Stroke Riskometer
  Interventions: Drug: Drug Capsule (Valsartan + Amlodipine + Rosuvastatin)
- Placebo + No Riskometer (Usual Care) (No Intervention): Participants will be randomized to use placebo polypill and will not use the Stroke Riskometer

INTERVENTIONS:
Drug: Drug Capsule (Valsartan + Amlodipine + Rosuvastatin) — Polypill with 3 medications (Valsartan 80 mg + Amlodipine 5 mg + Rosuvastatin 10 mg)
  Arms: Polypill + No Stroke Riskometer (Usual care); Polypill + Stroke Riskometer
Behavioral: Stroke Riskometer — Participants will be randomized to use Stroke Riskometer App for lifestyle modifications
  Arms: Placebo + Stroke Riskometer; Polypill + Stroke Riskometer

SUMMARY:
This study is a phase III, prospective, placebo-controlled randomized clinical trial involving 8,518 subjects with low to moderate stroke risk, followed for 3 years in Brazil. Participants will be randomized to receive either the polypill (valsartan 80 mg, amlodipine 5 mg, and rosuvastatin 10 mg), with dose adjustment of amlodipine to 2.5 mg for patients experiencing adverse events, or a placebo, and to either use the Stroke Riskometer for lifestyle modification or receive usual care. The purpose of the study is to test whether the polypill, alone or in combination with lifestyle modification, will reduce the incidence of stroke and cognitive impairment in this population.

DETAILED DESCRIPTION:
Background and Aims The increasing burden of stroke and dementia provides strong evidence that current primary prevention strategies are insufficient, as 80% of strokes occur in individuals with low to moderate risk. The purpose of this study is to test whether a polypill, used alone or in combination with lifestyle modification, will reduce the incidence of stroke and cognitive impairment in a population with low to moderate stroke risk.

Methods

This is a phase III, multicenter, prospective, double-blind, placebo-controlled randomized clinical trial of 8,518 subjects with low to moderate stroke risk, followed for 3 years. The study will include 80 Health Units affiliated with 20 research centers in Brazil. After a run-in phase (30 days, all participants with active drug), participants will be randomized to receive either the polypill (valsartan 80 mg, amlodipine 5 mg, and rosuvastatin 10 mg) or a placebo (with dose adjustment of amlodipine to 2.5 mg for patients experiencing adverse events), and to either use the Stroke Riskometer for lifestyle modification or receive usual care. It will be included: (1)adults aged 50-75 years; (2) no previous history of stroke, TIA or cardiovascular disease; (3)systolic blood pressure (BP) 121-139 mmHg; (4) one or more lifestyle risk factors (smoking, overweight, physical inactivity or inadequate diet. It will be excluded patients with hypercholesterolemia or diabetes or take other antihypertensive drugs or open label statins. Subjects will be randomized under a minimization process:

* Age: 50-64 vs 65-75
* Sex: men vs women
* BP: 121-130 vs 131-139
* Education level: <5 years vs > 5 years
* Total Cholesterol: <5 mmol (194 mg/dl) vs <5 mmol (194 mg/dl)

The study will be conducted in 2 parts:

Part 1. Family Health Strategy Units (10 clusters) located in Porto Alegre will be eligible to participate in part 1, which will assess surrogate endpoints in 370 patients included in the study in 9 months (blood pressure reduction and change in stroke risk by the scale LS7). Also we will evaluate the strategies, and barriers for implementation and adverse events.

Part 2. 80 Family Health Strategy Units, affiliated with 20 research centers, in the 5 Brazilian regions, 8,518 participants followed for 3 years measuring stroke incidence and cognitive decline rate as the primary outcome. Expected results in primary outcome: to reduce the incidence of stroke and cognitive decline in the group of polypill and / or polypill + Riskometer. Secondary outcome: to reduce stroke, MI and cardiovascular death.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 50-75 years;
* no previous history of stroke, TIA or cardiovascular disease;
* systolic blood pressure (SBP) 121-139 mmHg;
* with one or more lifestyle risk factors: smoking, overweight (BMI> 25 kg / m2), physical inactivity (WHO criteria for aerobic physical activity <150 minutes / week or at least 75 minutes of aerobic physical activity of vigorous intensity during the week or an equivalent combination of activity of moderate and vigorous intensity) or inadequate diet / poor eating habits (low intake of fruits and vegetables, fish, whole grains, high intake of drinks sweetened with sodium and sugar)
* owns or has access to a cell phone that can receive text messages.

Exclusion Criteria:

* Diagnostic of hypercholesterolemia (> 190mg/dL LDL cholesterol) or diabetes or take other antihypertensive drugs or open label statins;
* Contraindication to the medication
* Life expectancy < 5 years
* Participation in another clinical trial

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8518 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2029-12-14 (Estimated); Study Completion 2030-12-14 (Estimated)

PRIMARY OUTCOMES:
Stroke | 3 years
  Incidence of Ischemic or hemorrhagic stroke
Cognitive decline | 3 years
  Cognitive decline rate

SECONDARY OUTCOMES:
MACE | 3 years
  Incidence of Stroke/TIA, Myocardial infarction, hospitalization for cardiovascular cause and cardiovascular death comparing the polypill and placebo group and comparing riskometer and no riskometer group
Life's Essential 8 Score (LE8) | 3 years
  Difference of LE8 at the baseline and in 3 years comparing the 4 groups
Systolic blood pressure | 3 years
  Systolic blood pressure in 3 years comparing the 4 groups
Cholesterol | 3 years
  Total and LDL cholesterol in 3 years comparing the 4 groups
Numbers of Cardiovascular risk factors | 3 years
  Numbers of Cardiovascular risk factors in the riskometer group comparing to the usual care
Quality of Life Analysis | 3 years
  Quality of life analysis as measured by EuroQol/EQ5D comparing the 4 groups. The score range from 0.33 to 1 with higher scores indicating better quality if life
Life's Essential 8 Score (LE8) | 3 years
  Proportion of participants with decreased risk for LE8 comparing the 4 groups. The score range from 0 to 100 with higher scores indicating better cardiovascular health
Cost of stroke treatment | 3 years
  Cost of primary care in the primary care unit

CONTACTS AND LOCATIONS:
Overall Officials: Sheila CO Martins, PhD, Principal Investigator — Hospital Moinhos de Vento; Michael Brainin, MD, Study Chair — Danube University Krems, Austria; Valery Feigin, PhD, Study Chair — AUT University, Oakland, New Zealand; Thais L Secchi, MSc, Study Director — Hospital Moinhos de Vento
Locations (2):
- Brazil (2):
  - Unidade de Saúde Santa Cecília / Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul

REFERENCES:
- [Background] GBD 2015 Neurological Disorders Collaborator Group. Global, regional, and national burden of neurological disorders during 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet Neurol. 2017 Nov;16(11):877-897. doi: 10.1016/S1474-4422(17)30299-5. Epub 2017 Sep 17. PMID 28931491
- [Background] Feigin VL, Roth GA, Naghavi M, Parmar P, Krishnamurthi R, Chugh S, Mensah GA, Norrving B, Shiue I, Ng M, Estep K, Cercy K, Murray CJL, Forouzanfar MH; Global Burden of Diseases, Injuries and Risk Factors Study 2013 and Stroke Experts Writing Group. Global burden of stroke and risk factors in 188 countries, during 1990-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet Neurol. 2016 Aug;15(9):913-924. doi: 10.1016/S1474-4422(16)30073-4. Epub 2016 Jun 9. PMID 27291521
- [Background] The Lancet Neurology. The shared burden of stroke and dementia. Lancet Neurol. 2016 Aug;15(9):891. doi: 10.1016/S1474-4422(16)30132-6. No abstract available. PMID 27478943
- [Background] Feigin VL, Norrving B, George MG, Foltz JL, Roth GA, Mensah GA. Prevention of stroke: a strategic global imperative. Nat Rev Neurol. 2016 Sep;12(9):501-12. doi: 10.1038/nrneurol.2016.107. Epub 2016 Jul 22. PMID 27448185
- [Background] Forouzanfar MH, Liu P, Roth GA, Ng M, Biryukov S, Marczak L, Alexander L, Estep K, Hassen Abate K, Akinyemiju TF, Ali R, Alvis-Guzman N, Azzopardi P, Banerjee A, Barnighausen T, Basu A, Bekele T, Bennett DA, Biadgilign S, Catala-Lopez F, Feigin VL, Fernandes JC, Fischer F, Gebru AA, Gona P, Gupta R, Hankey GJ, Jonas JB, Judd SE, Khang YH, Khosravi A, Kim YJ, Kimokoti RW, Kokubo Y, Kolte D, Lopez A, Lotufo PA, Malekzadeh R, Melaku YA, Mensah GA, Misganaw A, Mokdad AH, Moran AE, Nawaz H, Neal B, Ngalesoni FN, Ohkubo T, Pourmalek F, Rafay A, Rai RK, Rojas-Rueda D, Sampson UK, Santos IS, Sawhney M, Schutte AE, Sepanlou SG, Shifa GT, Shiue I, Tedla BA, Thrift AG, Tonelli M, Truelsen T, Tsilimparis N, Ukwaja KN, Uthman OA, Vasankari T, Venketasubramanian N, Vlassov VV, Vos T, Westerman R, Yan LL, Yano Y, Yonemoto N, Zaki ME, Murray CJ. Global Burden of Hypertension and Systolic Blood Pressure of at Least 110 to 115 mm Hg, 1990-2015. JAMA. 2017 Jan 10;317(2):165-182. doi: 10.1001/jama.2016.19043. PMID 28097354
- [Background] Farzadfar F, Finucane MM, Danaei G, Pelizzari PM, Cowan MJ, Paciorek CJ, Singh GM, Lin JK, Stevens GA, Riley LM, Ezzati M; Global Burden of Metabolic Risk Factors of Chronic Diseases Collaborating Group (Cholesterol). National, regional, and global trends in serum total cholesterol since 1980: systematic analysis of health examination surveys and epidemiological studies with 321 country-years and 3.0 million participants. Lancet. 2011 Feb 12;377(9765):578-86. doi: 10.1016/S0140-6736(10)62038-7. Epub 2011 Feb 3. PMID 21295847
- [Background] O'Regan C, Wu P, Arora P, Perri D, Mills EJ. Statin therapy in stroke prevention: a meta-analysis involving 121,000 patients. Am J Med. 2008 Jan;121(1):24-33. doi: 10.1016/j.amjmed.2007.06.033. PMID 18187070
- [Background] Feigin VL, Norrving B, Mensah GA. Primary prevention of cardiovascular disease through population-wide motivational strategies: insights from using smartphones in stroke prevention. BMJ Glob Health. 2017 Apr 4;2(2):e000306. doi: 10.1136/bmjgh-2017-000306. eCollection 2016. PMID 28589034
- [Background] Yusuf S, Lonn E, Pais P, Bosch J, Lopez-Jaramillo P, Zhu J, Xavier D, Avezum A, Leiter LA, Piegas LS, Parkhomenko A, Keltai M, Keltai K, Sliwa K, Chazova I, Peters RJ, Held C, Yusoff K, Lewis BS, Jansky P, Khunti K, Toff WD, Reid CM, Varigos J, Accini JL, McKelvie R, Pogue J, Jung H, Liu L, Diaz R, Dans A, Dagenais G; HOPE-3 Investigators. Blood-Pressure and Cholesterol Lowering in Persons without Cardiovascular Disease. N Engl J Med. 2016 May 26;374(21):2032-43. doi: 10.1056/NEJMoa1600177. Epub 2016 Apr 2. PMID 27039945
- [Background] Brainin M, Feigin V, Martins S, Matz K, Roy J, Sandercock P, Teuschl Y, Tuomilehto J, Wiseman A. Cut stroke in half: Polypill for primary prevention in stroke. Int J Stroke. 2018 Aug;13(6):633-647. doi: 10.1177/1747493018761190. Epub 2018 Feb 20. PMID 29461155
- [Background] Elley CR, Gupta AK, Webster R, Selak V, Jun M, Patel A, Rodgers A, Thom S. The efficacy and tolerability of 'polypills': meta-analysis of randomised controlled trials. PLoS One. 2012;7(12):e52145. doi: 10.1371/journal.pone.0052145. Epub 2012 Dec 19. PMID 23284906
- [Background] Roshandel G, Khoshnia M, Poustchi H, Hemming K, Kamangar F, Gharavi A, Ostovaneh MR, Nateghi A, Majed M, Navabakhsh B, Merat S, Pourshams A, Nalini M, Malekzadeh F, Sadeghi M, Mohammadifard N, Sarrafzadegan N, Naemi-Tabiei M, Fazel A, Brennan P, Etemadi A, Boffetta P, Thomas N, Marshall T, Cheng KK, Malekzadeh R. Effectiveness of polypill for primary and secondary prevention of cardiovascular diseases (PolyIran): a pragmatic, cluster-randomised trial. Lancet. 2019 Aug 24;394(10199):672-683. doi: 10.1016/S0140-6736(19)31791-X. PMID 31448738
- [Background] Sung J, Jeong JO, Kwon SU, Won KH, Kim BJ, Cho BR, Kim MK, Lee S, Kim HJ, Lim SH, Park SW, Park JE. Valsartan 160 mg/Amlodipine 5 mg Combination Therapy versus Amlodipine 10 mg in Hypertensive Patients with Inadequate Response to Amlodipine 5 mg Monotherapy. Korean Circ J. 2016 Mar;46(2):222-8. doi: 10.4070/kcj.2016.46.2.222. Epub 2016 Mar 21. PMID 27014353
- [Background] Brainin M, Feigin V, Bath PM, Collantes E, Martins S, Pandian J, Sacco R, Teuschl Y. Multi-level community interventions for primary stroke prevention: A conceptual approach by the World Stroke Organization. Int J Stroke. 2019 Oct;14(8):818-825. doi: 10.1177/1747493019873706. Epub 2019 Sep 9. PMID 31500553
- [Background] Parmar P, Krishnamurthi R, Ikram MA, Hofman A, Mirza SS, Varakin Y, Kravchenko M, Piradov M, Thrift AG, Norrving B, Wang W, Mandal DK, Barker-Collo S, Sahathevan R, Davis S, Saposnik G, Kivipelto M, Sindi S, Bornstein NM, Giroud M, Bejot Y, Brainin M, Poulton R, Narayan KM, Correia M, Freire A, Kokubo Y, Wiebers D, Mensah G, BinDhim NF, Barber PA, Pandian JD, Hankey GJ, Mehndiratta MM, Azhagammal S, Ibrahim NM, Abbott M, Rush E, Hume P, Hussein T, Bhattacharjee R, Purohit M, Feigin VL; Stroke RiskometerTM Collaboration Writing Group. The Stroke Riskometer(TM) App: validation of a data collection tool and stroke risk predictor. Int J Stroke. 2015 Feb;10(2):231-44. doi: 10.1111/ijs.12411. Epub 2014 Dec 10. PMID 25491651
- [Background] Krishnamurthi R, Hale L, Barker-Collo S, Theadom A, Bhattacharjee R, George A, Arroll B, Ranta A, Waters D, Wilson D, Sandiford P, Gall S, Parmar P, Bennett D, Feigin V. Mobile Technology for Primary Stroke Prevention: A Proof-of-Concept Pilot Randomized Controlled Trial. Stroke. 2019 Jan;50(1):196-198. doi: 10.1161/STROKEAHA.118.023058. Epub 2018 Nov 21. PMID 30580699
- See also: The HEARTS technical package provides a strategic approach to improving cardiovascular health in countries. It comprises six modules and an implementation guide — https://www.who.int/publications/i/item/hearts-technical-package